CLINICAL TRIAL: NCT06694896
Title: Microarray Application in Newborns With Multiple Congenital Anomalies: Genotype-Phenotype Correlation
Brief Title: Microarray Application in Newborns With Multiple Congenital Anomalies
Acronym: CNV-MCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, RAMAZAN KEÇECİ, Principal Investigator (Specialist), Konya City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-006
Record Dates: First submitted 2024-11-10; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Multiple Abnormalies
Keywords: newborn; multipl congenital anomalies; microarray; copy number variant

STUDY DESIGN:
Intervention Model Description: Newborns with two major or one major and two minor, or three or more minor congenital anomalies were included. Microarray studies were performed on patients who met the inclusion criteria. CNVs identified were examined in relevant databases, and pathogenicity was assessed. Detected alterations were compared with the clinical findings in the patient database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MCA (Other): Multipl Congenital Anomalies
  Interventions: Diagnostic Test: Microarray Application

INTERVENTIONS:
Diagnostic Test: Microarray Application — Microarray studies were performed on patients who met the inclusion criteria. CNVs identified were examined in relevant databases, and pathogenicity was assessed. Detected alterations were compared with the clinical findings in the patient database.

SUMMARY:
Objective:

Congenital anomalies are defined as abnormalities of body structure or function that are present at birth and have developed prenatally. Microarray is considered the first-tier diagnostic test for patients with multiple congenital anomalies. The aim of this study is to determine the relationship between microarray results and the phenotype in newborns with multiple congenital anomalies, contribute to patient management by comparing with similar cases in the literature, detect previously unidentified Copy Number Variations (CNV), investigate the hereditary origin of the detected changes, and provide appropriate genetic counseling.

DETAILED DESCRIPTION:
Method:

Between December 2022 and November 2023, newborns with multiple congenital anomalies requiring follow-up and treatment in the Neonatal Intensive Care Unit of Konya City Hospital were evaluated. Newborns with examination findings suggesting a recognizable numerical chromosome anomaly or a history of teratogenicity were excluded from the study. Newborns with two major or one major and two minor, or three or more minor congenital anomalies were included. Microarray studies were performed on patients who met the inclusion criteria. CNVs identified were examined in relevant databases, and pathogenicity was assessed. Detected alterations were compared with the clinical findings in the patient database.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with two major or one major and two minor, or three or more minor congenital anomalies were included

Exclusion Criteria:

* Newborns with examination findings suggesting a recognizable numerical chromosome anomaly
* History of teratogenicity

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Copy Number Variant | 1 year
  Primary outcome variable: To investigate the relationship between chromosomal disorders and newborns with Multiple Congenital Anomalies

SECONDARY OUTCOMES:
Copy Number Variant | 1 year
  Secondary outcome variable: To investigate the relationship between parental transmission of chromosomal disorders found in newborns with Multiple Congenital Anomalies.

CONTACTS AND LOCATIONS:
Locations (1):
- Konya City Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the study is published, it can be made available to other researchers.

REFERENCES:
- [Background] Szczaluba K, Nowakowska B, Sobecka K, Smyk M, Castaneda J, Klapecki J, Kutkowska-Kazmierczak A, Smigiel R, Bocian E, Radkowski M, Demkow U. Application of Array Comparative Genomic Hybridization in Newborns with Multiple Congenital Anomalies. Adv Exp Med Biol. 2016;912:1-9. doi: 10.1007/5584_2016_235. PMID 26987320
- [Background] Szczaluba K, Demkow U. Array comparative genomic hybridization and genomic sequencing in the diagnostics of the causes of congenital anomalies. J Appl Genet. 2017 May;58(2):185-198. doi: 10.1007/s13353-016-0376-z. Epub 2016 Nov 18. PMID 27858254